CLINICAL TRIAL: NCT01430767
Title: Measuring Adherence to Standard-of-Care Medication for Depression and ADHD in a College Student Population
Brief Title: Measuring Adherence to Medication for Depression and Attention-deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: WFBMC-Psych-17564
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2015-12

CONDITIONS: Major Depressive Disorder; Attention-deficit Hyperactivity Disorder (ADHD)
Keywords: adherence
MeSH Terms: conditions — Depressive Disorder, Major; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Depression: Ten subjects with diagnosis of major depressive disorder from the Wake Forest University Student Health Clinic, being treated with FDA-approved standard-of-care medication for depression.
- ADHD: Ten subjects with a diagnosis of attention-deficit hyperactivity disorder (ADHD) from the Wake Forest University Student Health Clinic, being treated with FDA-approved standard-of-care medication for their ADHD.

SUMMARY:
Poor adherence is a common reason for treatment failure in many fields of medicine, and likely affects common psychiatric treatments as well. Members of the present study team have used Medication Event Monitoring System (MEMS®) caps effectively to objectively monitor adherence in skin disease, and have shown that they provide a much more accurate measure of adherence behavior than self-reports, pill counts, or serum drug concentrations. The present study will use MEMS® caps to measure adherence in 10 patients with depression and 10 patients with attention-deficit hyperactivity disorder (ADHD) from a student clinic population. The aims will be to show the usefulness of MEMS® caps in measuring adherence to psychiatric treatment, and gather data on typical adherence rates for depression and ADHD patients on typical treatment regimens. The data obtained will be used to inform future studies that use an intervention to improve adherence behavior and ultimately disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female, at least 18 years of age, using the Student Health Clinic, with a diagnosis of depression or ADHD.
* Written consent of participation must be given by the subject.

Exclusion Criteria:

* Subject is less than 18 years of age.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication while participating in the study. (Patients who are on a stable dose of non-study-related prescription medications for at least 4 weeks prior to the study, and throughout the study period, are not excluded.)
* Female patients whose medications may be harmful during pregnancy must be on an acceptable form of birth control, otherwise they will not be eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty male and female subjects, ten with depression and ten with ADHD, will be recruited. Subjects will be recruited from the Student Health Clinic at Wake Forest University, as we plan to assess adherence in a typical population of college students with depression or ADHD.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adherence to Standard-of-Care Medication for Depression or ADHD | 4 weeks
  Adherence to standard-of-care medication for depression or ADHD will be objectively measured using a bottle fitted with a Medication Event Monitoring System (MEMS®) cap and the percentage of prescribed doses taken will be reported as the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guy K Palmes, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States